CLINICAL TRIAL: NCT03627442
Title: Pilot Study: Post-operative Outcomes of Enhanced Energy Delivery Dissection for Mastectomy Breast Flap Creation With Immediate Breast Reconstruction
Brief Title: Post-op Outcomes of Enhanced Energy Delivery Dissection for Mastectomy With Immediate Breast Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Invuity, Inc. (Industry)
Collaborators: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-8737
Record Dates: First submitted 2018-07-18; First posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy

STUDY DESIGN:
Intervention Model Description: Single blinded, randomized controlled pilot study (n=15) Only breast surgeon knows which device was used for each breast at initiation of surgery
Masking Description: Initially, only breast surgeons knows which of the two devices was used for each breast, not plastic surgeon
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mastectomy with PhotonBlade (Active Comparator): Patients undergoing double mastectomy with immediate reconstruction with expanders. One breast will be randomly selected to be operated with PhotonBlade
  Interventions: Procedure: Mastectomy with PhotonBlade
- Mastectomy with Bovie (Active Comparator): Patients undergoing double mastectomy with immediate reconstruction with expanders. One breast will be randomly selected to be operated with Bovie.
  Interventions: Procedure: Mastectomy with Bovie

INTERVENTIONS:
Procedure: Mastectomy with PhotonBlade — One of the breasts of each patient undergoing double mastectomy will be randomly assigned to breast flap creation with PhotonBlade
  Arms: Mastectomy with PhotonBlade
Procedure: Mastectomy with Bovie — One of the breasts of each patient undergoing double mastectomy will be randomly assigned to breast flap creation with Bovie
  Arms: Mastectomy with Bovie

SUMMARY:
Principal Investigator: Sheldon Feldman, MD Co-Principal Investigator: Mohamad Sebai, MD Department of Surgery, Montefiore Medical Center - Einstein College of Medicine

Title Pilot Study: Post-operative outcomes of enhanced energy delivery dissection for mastectomy breast flap creation with immediate breast reconstruction Goal Determine the feasibility of a study design that includes the evaluation of breast flap viability, postoperative surgical site drainage, post-operative pain/surgical site complications, time to complete mastectomy with Photonblade (PB) vs traditional electrosurgery devices.

Overall outcome If determined feasible, consider going to clinical trial. Timing 6 months starting after execution of contract Study population Women between 18-65 years old Choose bilateral mastectomy followed by immediate breast reconstruction (through tissue expander insertion) No inflammatory breast cancer/no radiotherapy Study design Single blinded, randomized controlled pilot study (n=15) Only breast surgeon knows which device was used for each breast Study feasibility endpoints Flap Viability - compare perfusion, using PhotonVue, of flaps creation using PB vs Bovie (left is better, right is better or they are similar) Site drainage - Measure drainage volume and duration Pain scores and complications - Subjective pain assessment on days 1, 2, 3, 7 and 30 post-op. (Pain visual Analog Scale).

Surgical site complications will be recorded up to 30-days post-op. Time to completion of mastectomy flap using PB vs Bovie will be recorded. (Time in minutes between initial incision and completion of mastectomy for each side) Analysis Descriptive analysis will be performed to examine data distribution, missing data and data errors.

Continuous variables will be summarized using means or medians; categorical variables will be summarized using proportions.

CLINICAL TRIAL Objectives Determine if post-op flap viability differs between women getting mastectomy flap creation using PB vs Bovie Determine if post-op site drainage measures differs between two devices Determine if post-op pain measures differ when using PB vs Bovie Determine if time to mastectomy flap creation differs between using Bovie and PB

DETAILED DESCRIPTION:
Pilot Study: Post-Operative Outcomes of Enhanced Energy Delivery Dissection for Mastectomy Breast Flap Creation with Immediate Breast Reconstruction

Principal Investigator Sheldon M. Feldman, MD Chief, Division of Breast Surgery & Breast Surgical Oncology Director, Breast Cancer Services; Professor of Surgery Montefiore Medical Center- Albert Einstein College of Medicine New York, NY Email: sfeldman@montefiore.org

Co-Principal Investigator Mohamad E. Sebai, MD General Surgery Resident Montefiore Medical Center- Albert Einstein College of Medicine New York, NY Email: msebai@montefiore.org

Biostatistics: Michael Parides, PhD Professor Department of Surgery Montefiore Medical Center- Albert Einstein College of Medicine New York, NY Email: mparides@montefiore.org

Patricia Friedmann, MS Assistant Professor Department of Surgery Montefiore Medical Center- Albert Einstein College of Medicine New York, NY Email: patricia.friedmann@einstein.yu.edu

1. Rationale:

   Breast cancer is the second leading cause of cancer deaths among women in the United States. The American Cancer Society (ACS) estimated that 230,480 new cases of invasive breast cancer, a 19.8% increase over the ACS's 2009 estimates, and 39,520 deaths due to the disease would occur in 2011(1). In addition to breast conserving treatments, mastectomy can be an important and definitive treatment option for selected patients. Breast reconstruction has been shown to improve quality of life scores in patients treated with mastectomy (2). Immediate Breast reconstruction (IBR) after mastectomy has typically been performed using prosthetic devices or autologous tissue transplantation (3).

   Skin sparing mastectomy is a commonly used method of surgical treatment for breast cancer that allows for immediate breast reconstruction (4). Preservation of the breast skin envelope (breast flap) provides excellent cosmetic results and the overall sensation is largely maintained (4-7). An important factor for breast reconstruction success is the creation of a well perfused breast flap, with minimum flap injury (8-10). One of the major complications associated with this surgery is breast flap death (necrosis, 11). This complication then requires the patient to endure further operations, prolonged hospital stays, and higher hospital costs. Rates of native skin flap ischemia and necrosis after skin-sparing mastectomy vary from 2% to 30% (11,12). Some evidence suggests that this flap necrosis could be due to decreased or loss of viability/ blood supply (ischemia) as a result of the thermal injury caused by traditional dissection devices (Bovie cautery) use for breast flap creation (13). The use of traditional dissection devices remains to be the most common in creating breast flaps, despite how old this technology is. Newer dissection devices that uses modern technology for enhanced energy delivery has been introduced recently, however, there is still paucity of data in regards to the clinical outcomes of using these devices for the cases of mastectomy and IBR.

   PhotonBlade (Invuity, San Francisco, CA, USA) has been approved by United States Food and Drug Administration (FDA). PhotonBlade is a dynamic precision illuminator with enhanced energy delivery dissection device. The dynamic precision illumination is a thermally cool illumination technology that allows a uniformal illumination without glare or shadow (14). The enhanced energy delivery technology allows low thermal spread, surgeon controlled edge temperature, and wet field use (14). As such, PhotonBlade allows better blade control for achieving adequate visualization, hemostasis, with a minimum collateral damage to the created flap. The use of PhotonBlade demonstrated the least penetrating thermal tissue damage/spread when compared to other modern dissection devices (Valleylab Pencil, Valleylab EDGE Coated Pencil, PlasmaBlade 3.0S and PlasmaBlade 4.0)(15).

   The aim of this pilot study is to evaluate the feasibility of measuring breast flap viability, postoperative surgical site drainage, post-operative pain/ surgical site complications, and time to complete mastectomy with the use of enhanced energy delivery dissection devices, PhotonBlade, in comparison to traditional electrosurgery devices.
2. Study Design:

   This is a single-blinded, controlled pilot study (n=15) to determine the feasibility of comparing postoperative flap viability and surgical site drainage between patients randomized to breast flap creation by PhotonBlade on one breast and by a Bovie cautery (Control) for the contralateral breast. Candidates will have elected to undergo bilateral post-mastectomy IBR through tissue expander insertion. Participants meeting inclusion criteria will be enrolled and baseline data collection completed prior to randomization and surgery.

   Patients will be blinded in regards to which side will be treated with which cautery device. Initially, the plastic surgeon will be blinded as to the electrocautery device used on the breast until after completing the flap evaluation, when the plastic surgeon will be unblinded. This is done to allow the plastic surgeon to use same dissection device for each breast side during the reconstruction part of the surgery. Only the breast oncology surgeon has initial knowledge of which device was used for each breast flap. Patient-specific surgical details will be recorded intraoperatively. Following the surgery, post-operative flap perfusion will be recorded using PhotonVue imaging system and will be used a tool for flap viability assessment by the plastic surgeon clinical evaluation. Surgical site drainage will be measured until drainage removal. Post- operative pain scores and the occurrence of adverse events will be recorded up until 30 days post-op. Before starting enrollment, the breast and plastic surgeons will do up to 5 non-pilot study cases using PhotonBlade in order be familiar with the device. Figure 1 demonstrates study design schema for the pilot study. Figure 1 does not include the up to 5 non-pilot study cases.
3. Sample Size:

   The proposed sample size of 15 patients for this pilot study is based on ensuring acceptable operating characteristics for the decision process for assessing feasibility. Feasibility will be determined by whether breast flaps created using the PhotonBlade have better viability than those created using Bovie cautery. The null hypothesis is that the probability that flaps created using the PhotonBlade have better viability than those created by Bovie cautery (π) is less than one-half. The alternative hypothesis is that this probability is greater than one-half. Feasibility is defined as observing superior viability with the PhotonBlade in 10 or more of the 15 randomized patients. The sample size of 15 ensures that the false positive rate (Type I error) for determining feasibility using this definition is 0.15 (i.e., the binomial probability of observing 10 or more patients with better viability using the PhotonBlade out of 15 total patients given π=0.50 is 0.15). This probability (i.e., power) is 0.85 under the alternative that π=0.75, and 0.72 under the alternative that π=0.70.
4. Randomizations:

   Patients will have their breasts randomized, with the left breast receiving mastectomy flap creation using the randomized assignment (PhotonBlade or Bovie cautery), and the right breast receiving the other approach. Randomization of breast side will be performed by the breast surgical oncologist on the day of the surgery from a master randomization list created by the study statistician. A simple randomization scheme will be employed.
5. Flap Perfusion Viability This will be done by the plastic surgeon who will evaluate the flaps by using PhotonVue near-infrared fluorescence images for flap perfusion of each breast flap after the mastectomy and before the immediate breast reconstruction.

   PhotonVue is an FDA approved fluorescence imaging system that is used as an adjuvant assessment tool of tissue perfusion, and blood circulation of free flaps used in plastic, micro- reconstruction, and organ transplant surgeries.16 PhotonVue images of the flap perfusion will be taken at 45-60 seconds post ICG injection.

   For each case, the plastic surgeons will report one of three outcomes: a) Left breast flap has a better viability, b) Right breast flap has a better viability, or c) both sides are similarly viable. After unbinding, the results will be reported according to the usage of PhotonBlade or Bovie cautery for each side.
6. Surgical Site Drainage Assessments This will be done by measuring surgical site drainage volume and days until removal of the drains for each breast.
7. Post-Operative Pain Assessment Pain Visual Analog Scale will be used to assess pain preoperatively and postoperatively. Patient will be asked to report their pain score for each breast using the validated Pain Visual Analog Scale (Appendix A). Short term post pain will be reported as the mean of pain scores up to day 7, and longer term post op pain will be the pain score at day 30 post op. Up to 30 days post-op follow-up medical records will be used to collect incidences of post op surgical site complications. Additionally, patients will be asked to report their experience at the 30 days follow up appointment. Their response will be recorded. They will be also asked to report one of the following: 1) I believe the right breast had a better patient reported outcomes based on my experience, 2) I believe the left breast had a better patient reported outcomes based on my experience, or 3) I believe both breasts had similar patient reported outcomes based on my experience. After completion of data collection of the 30 days post-op follow up visit, patients will be unblinded and they will be made aware of which dissection device was used for which breast.
8. Time for Mastectomy Completion This will be done by measuring time in minutes from the incision time until the completion of mastectomy for each breast side.
9. Outcome Evaluation:

   Sources of data: The sources of the data are our institutional medical records system.

   Data collection: Data will be collected from the medical records through chart review process done by study team officials.

   Data analysis: The main analytic goal of this pilot study is assessment of feasibility which is based on the number of patients with PhotonBlade flaps having better viability than Bovie flaps (a "success"), and quantified by the exact (binomial) probability of observing at least that many successes if the true success probability is 0.5. Additional outcomes will be summarized numerically using descriptive statistics (appropriate point and interval estimates) and graphically (histograms, box-plots, stem and leaf plots as required).
10. Toxicity grading:

    All adverse events will be recorded and reported in accordance to The National Cancer Institute's published Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
11. Data Storage All study data will be stored within a password secured electronic dataset. Study data will be accessed only by IRB approved study staff.
12. Timeline:

The estimated period for the feasibility pilot study (n=15) is 6 months starting from signing the contract. Once IRB approval is attained for the pilot study, patient enrollment will begin. Patients data and study outcomes will be collected on rolling basis in parallel with patient enrollment and study execution. Once all data are gathered, data reporting will be done.

ELIGIBILITY:
Inclusion Criteria:

* Patients with or without breast cancer whom are candidates for and choose bilateral mastectomy followed by immediate breast reconstruction (tissue expander based breast reconstruction).
* Patients who had neoadjuvant chemotherapy are not excluded from participation
* Understand the study purpose, requirements, and risks.
* Be able and willing to give informed consent.

Exclusion Criteria:

* Inflammatory breast cancer
* Connective tissue disease
* Previous breast radiotherapy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-08-15 (Estimated); Primary Completion 2019-08-15 (Estimated); Study Completion 2019-10-15 (Estimated)

PRIMARY OUTCOMES:
Flap perfusion viability | Immediately after mastectomy
  This will be done by the plastic surgeon who will evaluate the flaps using PhotonVue images for flap perfusion of each breast flap after the mastectomy and before the immediate breast reconstruction.
  PhotonVue is an FDA approved fluorescence imaging system that is used as an adjuvant assessment tool of tissue perfusion, and blood circulation of free flaps used in plastic, micro- reconstruction, and organ transplant surgeries.16 PhotonVue images of the flap perfusion will be taken at 45-60 seconds post ICG injection.
  For each case, the plastic surgeons will report one of three outcomes: a) Left breast flap has a better viability, b) Right breast flap has a better viability, or c) both sides are similarly viable. After unbinding, the results will be reported according to the usage of PhotonBlade or Bovie cautery for each side.
Change in Surgical Site Drainage | Post surgery until removal of drains from each breast, assessed up to 5 weeks
  This will be done by measuring surgical site drainage volume until removal of the drains for each breast.
Post-Operative Pain Assessment | Change in pain for each breast will be assessed preoperatively and then postoperatively on days 1, 2, 3, 7 and 30.
  Pain Visual Analog Scale will be used to assess pain pre-operatively and post-operatively. Patient will be asked to report their pain score for each breast using the validated Pain Visual Analog Scale. The Visual Analog Scale For pain, asks the patient to draw a line indicating their level of pain on a 10 cm vertical line (where the bottom of the vertical line indicates no pain and the top indicates highest pain level). The line drawn by the patient will provide the pain score which will be calculated as the distance in mm from the bottom (no pain) level to the patient mark. As such, higher values will mean higher level of pain. Short term post pain will be reported as the mean of pain scores up to day 7, and longer term post op pain will be the pain score at day 30 post op. Up to 30 days post-op follow-up medical records will be used to collect incidences of post op surgical site complications.
Surgical Site Complications | Day 1, 2 and 3 pot-surgery (until discharge) and up to 30 days.
  Will document any surgical site complications.
Surgical Site Drainage - Time | Postsurgery and until removal of the drains
  This will be done by counting the days until removal of the drains for each breast

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Sebai, MD, Principal Investigator — Montefiore Medical Center; Sheldon Feldman, MD, Principal Investigator — Montefiore Medical Center

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] ACS. Breast Cancer Facts and Figures 2011-2012. (2012).
- [Background] Girotto JA, Schreiber J, Nahabedian MY. Breast reconstruction in the elderly: preserving excellent quality of life. Ann Plast Surg. 2003 Jun;50(6):572-8. doi: 10.1097/01.SAP.0000069064.68579.19. PMID 12783001
- [Background] Albornoz CR, Bach PB, Mehrara BJ, Disa JJ, Pusic AL, McCarthy CM, Cordeiro PG, Matros E. A paradigm shift in U.S. Breast reconstruction: increasing implant rates. Plast Reconstr Surg. 2013 Jan;131(1):15-23. doi: 10.1097/PRS.0b013e3182729cde. PMID 23271515
- [Background] Gonzalez EG, Rancati AO. Skin-sparing mastectomy. Gland Surg. 2015 Dec;4(6):541-53. doi: 10.3978/j.issn.2227-684X.2015.04.21. PMID 26645008
- [Background] Cho JW, Yoon ES, You HJ, Kim HS, Lee BI, Park SH. Nipple-Areola Complex Necrosis after Nipple-Sparing Mastectomy with Immediate Autologous Breast Reconstruction. Arch Plast Surg. 2015 Sep;42(5):601-7. doi: 10.5999/aps.2015.42.5.601. Epub 2015 Sep 15. PMID 26430632
- [Background] Martinez CA, Reis SM, Sato EA, Boutros SG. The Nipple-Areola Preserving Mastectomy: A Multistage Procedure Aiming to Improve Reconstructive Outcomes following Mastectomy. Plast Reconstr Surg Glob Open. 2015 Oct 20;3(10):e538. doi: 10.1097/GOX.0000000000000516. eCollection 2015 Oct. PMID 26579344
- [Background] van Verschuer VM, Maijers MC, van Deurzen CH, Koppert LB. Oncological safety of prophylactic breast surgery: skin-sparing and nipple-sparing versus total mastectomy. Gland Surg. 2015 Dec;4(6):467-75. doi: 10.3978/j.issn.2227-684X.2015.02.01. PMID 26645001
- [Background] Tindholdt TT, Saidian S, Tonseth KA. Microcirculatory evaluation of deep inferior epigastric artery perforator flaps with laser Doppler perfusion imaging in breast reconstruction. J Plast Surg Hand Surg. 2011 Jun;45(3):143-7. doi: 10.3109/2000656X.2011.579721. PMID 21682611
- [Background] Lin SJ, Nguyen MD, Chen C, Colakoglu S, Curtis MS, Tobias AM, Lee BT. Tissue oximetry monitoring in microsurgical breast reconstruction decreases flap loss and improves rate of flap salvage. Plast Reconstr Surg. 2011 Mar;127(3):1080-1085. doi: 10.1097/PRS.0b013e31820436cb. PMID 21364410
- [Background] Garvey PB, Salavati S, Feng L, Butler CE. Perfusion-related complications are similar for DIEP and muscle-sparing free TRAM flaps harvested on medial or lateral deep inferior epigastric Artery branch perforators for breast reconstruction. Plast Reconstr Surg. 2011 Dec;128(6):581e-589e. doi: 10.1097/PRS.0b013e318230c122. PMID 22094755
- [Background] Chirappapha P, Petit JY, Rietjens M, De Lorenzi F, Garusi C, Martella S, Barbieri B, Gottardi A, Andrea M, Giuseppe L, Hamza A, Lohsiriwat V. Nipple sparing mastectomy: does breast morphological factor related to necrotic complications? Plast Reconstr Surg Glob Open. 2014 Feb 7;2(1):e99. doi: 10.1097/GOX.0000000000000038. eCollection 2014 Jan. PMID 25289296
- [Background] Patel KM, Hill LM, Gatti ME, Nahabedian MY. Management of massive mastectomy skin flap necrosis following autologous breast reconstruction. Ann Plast Surg. 2012 Aug;69(2):139-44. doi: 10.1097/SAP.0b013e3182250e23. PMID 21734543
- [Background] Rusby JE, Smith BL, Gui GP. Nipple-sparing mastectomy. Br J Surg. 2010 Mar;97(3):305-16. doi: 10.1002/bjs.6970. PMID 20101646